CLINICAL TRIAL: NCT03293017
Title: Baclofen Bij de Behandeling Van Acute Alcoholontwenning
Brief Title: Baclofen in Managing Acute Alcohol Withdrawal
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22112015
Record Dates: First submitted 2017-06-19; First posted 2017-09-26 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2020-11

CONDITIONS: Alcohol Use Disorder; Alcohol Withdrawal
MeSH Terms: conditions — Alcoholism | interventions — Diazepam; Baclofen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baclofen 30 mg/day (Experimental): baclofen 30 mg/day
  Interventions: Drug: Diazepam 10 MG; Drug: Baclofen 30mg
- Baclofen 60 mg/day (Experimental)
  Interventions: Drug: Diazepam 10 MG; Drug: Baclofen 60mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Diazepam 10 MG

INTERVENTIONS:
Drug: Diazepam 10 MG — If a patient's linical Institute Withdrawal Assessment (CIWA-ar) is more than 15 and did not decrease with 4 points compared to the previous score, they will be given oral diazepam to supress their symptoms, in a tablet of 10 mg.
Drug: Baclofen 30mg — Baclofen 30 mg/day given over three gifts daily
  Arms: Baclofen 30 mg/day
Drug: Baclofen 60mg — Baclofen 60 mg/day given over three gifts daily
  Arms: Baclofen 60 mg/day

SUMMARY:
The study goal is to investigate whether administration of oral baclofen forms an adequate treatment option in the management of acute alcohol withdrawal. The investigators will compare placebo with doses of baclofen 30 and 60 milligram per day (mg/day) in a randomized controlled trial including patients receiving symptom triggered diazepam.

DETAILED DESCRIPTION:
The conducted study will be randomized and single-blind (patients). After signing informed consent, the participants will be randomized in one of three groups: - placebo - baclofen 30 mg/day - baclofen 60 mg/day. The participants will be given a first administration after which the participant can receive Clinical Institute Withdrawal Assessment (CIWA-ar) score triggered diazepam, frequently assessed for at least 7 days. The primary outcome measure is the number of participants who received additional diazepam during these 7 days. The secondary outcome measure is the amount of diazepam received per group.

ELIGIBILITY:
Inclusion Criteria:

* Be an inpatient at the Psychiatry unit at UZBrussel at time of study enrollment.
* Be able to sign informed consent.
* Be male/female aged 18-60
* Primary diagnosis of alcohol use disorder.

Exclusion Criteria:

* Pregnancy and breastfeeding.
* Benzodiazepine use of more than the equivalent of diazepam 25 mg /day.
* Psychosis, confusion and acute mania.
* Parkinson's disease.
* Use of tricyclic antidepressants.
* Use of opioids.
* Known baclofen or benzodiazepine sensitivity or allergy.
* Unable to take oral medication.
* epidermal growth factor receptor (EGFR) < 60 (blood samples are routinely performed at intake).
* Prior diagnosis of epilepsy.
* Lactose intolerance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Need for additional diazepam | Measured 7 days after the start of alcohol withdrawal
  Amount of patients who lack the need of additional diazepam during 7-day alcohol withdrawal

SECONDARY OUTCOMES:
Dosage of additional diazepam needed | Measured 7 days after the start of alcohol withdrawal
  The difference between the total dosages of additional diazepam needed between the three study arms

CONTACTS AND LOCATIONS:
Overall Officials: Frieda Matthys, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- University Hospital Brussels, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided